CLINICAL TRIAL: NCT03191513
Title: The Acute Effects of Interesterification of Commercially Used Fats on Postprandial Fat Metabolism
Acronym: INTERMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HR-16/17-4397
Record Dates: First submitted 2017-05-23; First posted 2017-06-19 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2017-05

CONDITIONS: Healthy Adults; Postmenopausal Women
Keywords: Interesterified; Postprandial; Lipid
MeSH Terms: interventions — Rapeseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interesterified (Experimental): Interesterified blend of palm kernal and plam stearin. 50g fat.
  Interventions: Dietary Supplement: Interesterified blend of palm kernal and plam stearin
- Un-interesterified (Active Comparator): Un-interesterified blend of palm kernal and plam stearin. 50g fat.
  Interventions: Dietary Supplement: Un-interesterified blend of palm kernal and plam stearin
- Control (Active Comparator): Rapeseed oil. 50g fat.
  Interventions: Dietary Supplement: Rapeseed oil

INTERVENTIONS:
Dietary Supplement: Interesterified blend of palm kernal and plam stearin — 50 g fat provided as interesterified palm kernal and palm sterin blend in a single meal (sub-group, n=12, also have 75 mg 13C labelled tripalmatin and 1.2 g / kg body water deuterated water)
  Other Names: Interesterified blend
  Arms: Interesterified
Dietary Supplement: Un-interesterified blend of palm kernal and plam stearin — 50 g fat provided as un-interesterified palm kernal and palm sterin blend in a single meal (sub-group, n=12, also have 75 mg 13C labelled tripalmatin and 1.2 g / kg body water deuterated water)
  Other Names: Un-interesterified blend
  Arms: Un-interesterified
Dietary Supplement: Rapeseed oil — 50 g fat provided as rapeseed oil in a single meal (sub-group, n=12, also have 75 mg 13C labelled tripalmatin and 1.2 g / kg body water deuterated water)
  Other Names: Control fat
  Arms: Control

SUMMARY:
The purpose of this study is to investigate whether there are differences in postprandial metabolic indices following interesterified fats used commercially versus the corresponding un-interesterified blend.

DETAILED DESCRIPTION:
Aim: The current study aims to investigate the acute effects of commercially relevant interesterified 'hardstock' versus the corresponding un-interesterified blend on 8 h postprandial fat metabolism.

Hypothesis: Interesterification of a palm kernel and palm stearin fat blend, to produce a fat with a higher proportion of palmitic acid in the middle position of the triglyceride (TAG; but the same fatty acid composition), will alter postprandial lipid metabolism.

Subjects: Participants will include 24 healthy male and female (postmenopausal) volunteers aged between the ages of 45 and 75 years (since during this age metabolic changes start to take place).

Power calculation: Based on previous studies carried out by our group at King's College London, a sample size of 10 males and 10 females is required to detect a (clinically relevant) difference (for males and females separately) between means of 0.3 mmol/L maximal difference in 8 h plasma TAG concentration (standard deviation 0.33 mmol/L, significance level (alpha) of 0.05 and 80% power). 12 males and 12 females will be recruited to allow for a 20% drop out rate.

Expected value:The study will provide novel information on the acute effects of commercially relevant processed fats on postprandial lipaemia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 45-75 years
* Healthy (free of diagnosed diseases listed in exclusion criteria)
* Able to understand the information sheet and willing to comply with study protocol
* Able to give informed consent

Exclusion Criteria:

* Medical history of myocardial infarction, angina, thrombosis, stroke, cancer, liver or bowel disease or diabetes
* Body mass index < 20 kg/m2 or > 35 kg/m2
* Plasma cholesterol ≥7.5 mmol/L
* Plasma triacylglycerol > 3 mmol/L
* Plasma glucose > 7 mmol/L
* Blood pressure ≥140/90 mmHg
* Current use of antihypertensive or lipid lowering medications
* Premenopausal (for women)
* Alcohol intake exceeding a moderate intake (> 28 units per week)
* Current cigarette smoker (or quit withint the last 6 months)
* ≥ 20% 10-year risk of CVD as calculated using a risk calculator

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-27 (Actual)

PRIMARY OUTCOMES:
Area under plasma TAG concentration/ time curve | Up to 8 hours
  Postprandial area under plasma TAG concentration/ time curve

SECONDARY OUTCOMES:
Postprandial lipaemic response | Up to 8 hours
  Postprandial plamsa total fatty acid composition and non esterifed fatty acid
Positional composition retention (chylomicron) | Up to 6 hours
  Postprandial chylomicron TAG concentration and composition, TAG sn-2 fatty acid composition, total protein, apoB100 and apoB48

OTHER OUTCOMES:
Isotope lablelled parameters | Up to 8 hours
  In sub-group, n=12, postprandial 13C TAG concentration and breath CO2 13C
Lipoprotein particle size and number | Up to 8 hours
  Lipoprotein size (LDL, VLDL and HDL) and composition (total and small LDL, large VLDL and total and large HDL) measured by NMR
2 and 3 MCPD and glycidyl esters | Up to 8 hours
  Postprandial plasma 2 and 3-monochloropropane-1,2-diol or 3-chloropropane-1,2-diol glycidyl esters

CONTACTS AND LOCATIONS:
Overall Officials: Sarah EE Berry, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burnap SA, Sattler K, Pechlaner R, Duregotti E, Lu R, Theofilatos K, Takov K, Heusch G, Tsimikas S, Fernandez-Hernando C, Berry SE, Hall WL, Notdurfter M, Rungger G, Paulweber B, Willeit J, Kiechl S, Levkau B, Mayr M. PCSK9 Activity Is Potentiated Through HDL Binding. Circ Res. 2021 Nov 12;129(11):1039-1053. doi: 10.1161/CIRCRESAHA.121.319272. Epub 2021 Oct 4. PMID 34601896